CLINICAL TRIAL: NCT02372175
Title: Phase One, Open Label, Assessment of a Dengue-1-Virus-Live Virus Human Challenge - (DENV-1-LVHC) Virus Strain
Brief Title: Assessment of a Dengue-1-Virus-Live Virus Human Challenge - (DENV-1-LVHC) Virus Strain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S-14-09
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Dengue
Keywords: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose DENV-1-LVHC (Experimental): Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC) single low dose (0.5 mL of 6.5 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC)
- Medium dose DENV-1-LVHC (Experimental): Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC) single medium dose (0.5 mL of 6.5 x 10^4 PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC)
- High dose DENV-1-LVHC (Experimental): Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC) single high dose (0.5 mL of 6.5 x 10^5 PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC)

INTERVENTIONS:
Biological: Dengue-1 Virus-Live Virus Human Challenge (DENV-1-LVHC) — Dengue subtype 1 Challenge Virus (DENV-1) strain 45AZ5 administered as a single injection.

SUMMARY:
To evaluate the effectiveness of candidate dengue vaccine formulations, it is prudent to develop an appropriate challenge model. To this end, this first-in-human study will examine the safety and effectiveness of the Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) product and assess the ability of this virus strain to elicit an uncomplicated dengue-like illness.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or non-pregnant, non-lactating female
2. Age 18-45
3. Ability and willingness to sign informed consent
4. Passing score on comprehension test would be 75%, with up to 3 attempts
5. Available for the study period
6. Willing to use contraception for the duration of the study.
7. Provide consent for release of medical history records from primary care physician, college or university, urgent care or emergency room visit

Exclusion Criteria:

1. Female: pregnant or lactating
2. Heavy menstrual bleeding within the last 6 months-menstrual periods lasting longer than 6 days, or requiring 5 or more pads or tampons per day.
3. Female subjects using an intrauterine device (IUD) or Mirena®
4. Female subjects with fibroids or uterine polyps, endometriosis, dysmenorrhea, adenomyosis, and uterine scarring (e.g. after D&C)
5. Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B surface antigen, or flavi viruses (FV) to include dengue fever, West Nile, Yellow Fever, and Japanese encephalitis.
6. Diabetes, chronic obstructive pulmonary disease (COPD), peptic ulcer disease (PUD), or coronary artery disease (CAD)
7. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
8. Immediate family member (e.g. parent, sibling, child) with current, or a history of immunodeficiency or autoimmune disease
9. Current or a history of auto-immune disease
10. History of Guillain Barré syndrome (GBS)
11. Any history of FV infection or FV vaccination; or planned FV vaccination, outside the study protocol, during the study period
12. History of Bipolar Disorder, Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the subject from participating in the study.
13. Planned travel during the study period (180 days) which would interfere with the ability to complete all study visits
14. Recent (in the past 4 weeks) travel to any dengue endemic area. These potential subjects may be eligible for enrollment a minimum of 4 weeks later
15. Any laboratory abnormalities in the tests specified in Table 19 and Table 20 of the protocol. Note: these laboratory tests can be repeated if the screening physician believes 1) it is thought to be a normal variant of a healthy state or 2) it is a suspected laboratory error
16. Significant screening physical examination abnormalities at the discretion of the investigator
17. Women who intend to become pregnant or men who intend to father a child during the study period (approximately 6 months)
18. Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous vaccination or an allergy to specific medications/animals for which antigens may be in the virus preparations to include: shellfish allergy, fetal bovine serum, L-glutamine, neomycin and streptomycin
19. Planning to donate blood in the 1 year following inoculation with dengue
20. Participation or planned participation in another vaccine, drug, medical device, or medical procedure clinical trial in the 4 weeks prior to this trial, during the trial, or 6 months following inoculation in this clinical trial
21. Beliefs that bar the administration of blood products or transfusions
22. Positive urine screen for cocaine, amphetamines, or opiates
23. Currently taking Methadone or Suboxone
24. Currently taking anti-coagulant medication, aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
25. Chronic migraine headaches, defined as more than 15 headache days per month over a 3 month period of which more than 8 are migrainous, in the absence of medication over use
26. Chronic medical condition that, in the opinion of the investigator impacts subject safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10; Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Number of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Intensity of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Duration of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Occurrence of Solicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Intensity of Solicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Duration of Solicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Occurrence of unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Intensity of Unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Duration of Unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Occurrence of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Intensity of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Duration of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Occurrence of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Intensity of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Duration of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Number of Serious Adverse Events | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
Number of Serious Adverse Events | 6 months post virus inoculation

SECONDARY OUTCOMES:
Incubation period before onset of fever | Up to 28 days post virus inoculation
Viremia by Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) | Up to 28 days post virus inoculation
Occurrence of fever without other identifiable cause, such as strep throat or influenza | Up to 28 days post virus inoculation
  The occurrence of fever defined as greater than or equal to 38°C (100.4° F) measured at least 2 times in 24 hours but not lasting more than 96 hours up to 28 days post virus inoculation without other identifiable cause, such as strep infection or influenza.
Occurrence of Headache | Up to 28 days post virus inoculation
Grade of Headache | Up to 28 days post virus inoculation
Occurrence of Myalgia | Up to 28 days post virus inoculation
Grade of Myalgia | Up to 28 days post virus inoculation
Occurrence of Rash | Up to 28 days post virus inoculation
Grade of Rash | Up to 28 days post virus inoculation
Occurrence of Liver Function Tests Abnormalities [alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] | Up to 28 days post virus inoculation
Grade of Liver Function Tests Abnormalities [alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] | Up to 28 days post virus inoculation
Occurrence of Leukopenia | Up to 28 days post virus inoculation
Grade of Leukopenia | Up to 28 days post virus inoculation
Occurrence of Thrombocytopenia | Up to 28 days post virus inoculation
Grade of Thrombocytopenia | Up to 28 days post virus inoculation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Endy, MD, MPH, Principal Investigator — State University of New York, Upstate Medical University (SUNY-UMU)
Locations (1):
- State University of New York, Upstate Medical University (SUNY-UMU), Syracuse, New York, United States

REFERENCES:
- [Derived] Endy TP, Wang D, Polhemus ME, Jarman RG, Jasper LE, Gromowski G, Lin L, De La Barra RA, Friberg H, Currier JR, Abbott M, Ware L, Klick M, Paolino KM, Blair DC, Eckels K, Rutvisuttinunt W, Thomas SJ. A Phase 1, Open-Label Assessment of a Dengue Virus-1 Live Virus Human Challenge Strain. J Infect Dis. 2021 Feb 3;223(2):258-267. doi: 10.1093/infdis/jiaa351. PMID 32572470